CLINICAL TRIAL: NCT05251909
Title: A Multi-center, Randomized, Double-blind, Parallel-group, Placebo-controlled 3-Part Phase 3 Study to Demonstrate the Efficacy and Safety of Benralizumab in Patients With Eosinophilic Gastritis and/or Gastroenteritis (The HUDSON GI Study)
Brief Title: Efficacy and Safety of Benralizumab in Patients With Eosinophilic Gastritis and/or Gastroenteritis (The HUDSON GI Study)
Acronym: HUDSON GI
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated by the Sponsor based on emerging evidence in the pathology of eosinophilic upper gastrointestinal diseases. Recruitment for the study was terminated and only a small number of patients were recruited.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D3258C00001; 2021-000085-14 (EudraCT Number)
Record Dates: First submitted 2021-08-06; First posted 2022-02-23 (Actual); Results first posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Eosinophilic Gastritis; Eosinophilic Gastroenteritis
Keywords: Benralizumab; Eosinophilic Gastritis; Gastroenteritis; Intestinal Diseases; Stomach Diseases; Gastrointestinal Diseases; Digestive System Diseases
MeSH Terms: conditions — Eosinophilic enteropathy; Gastroenteritis; Intestinal Diseases; Stomach Diseases; Gastrointestinal Diseases; Digestive System Diseases | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a parallel-group efficacy and safety study with 2 arms that are participant and investigator blinded, with an open-label extension.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Benralizumab (Experimental): This arm is a subcutaneous dose of Benralizumab
  Interventions: Biological: Benralizumab
- Placebo (Placebo Comparator): This arm is a subcutaneous dose of Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Benralizumab — Benralizumab is a humanized, afucosylated, monoclonal antibody that binds specifically to the IL-5Rα on the target cell and thus directly depletes eosinophils through antibody-dependent cell-mediated cytotoxicity. Benralizumab has been widely approved for treatment of asthma.
  Other Names: Fasenra
  Arms: Benralizumab
Biological: Placebo — Placebo will be injected as a comparator to injection with Benralizumab to examine effect on both the signs and symptoms of EG/EGE and the underlying eosinophilic inflammation, with dual primary outcome variables
  Arms: Placebo

SUMMARY:
This is a 3-part study. Part A is randomized, double-blinded, placebo-controlled and includes patients with eosinophilic gastritis and/or duodenal-only disease. After completing Part A, participants can continue to Part C - open-label benralizumab treatment period. Following the decision to close enrollment, patients in both Part A and Part C will be given the option to proceed to 6-months of open-label benralizumab treatment in Part D.

ELIGIBILITY:
Inclusion criteria:

* Aged >= 12 years of age at the time of signing the ICF or informed consent or assent form.
* Confirmed diagnosis of EG/EGE for at least 3 months prior to screening.
* Baseline Eosinophilic gastritis, with or without duodenitis, or eosinophilic duodenitis alone confirmed by biopsy with a gastric count of ≥30 eosinophils/hpf in at least 5 hpfs and/or duodenal eosinophil count ≥30 eosinophils/hpf in at least 3 hpfs without any other cause for the gastrointestinal eosinophilia.
* Symptoms including at least moderate abdominal pain, nausea, bloating, early satiety, and/or loss of appetite
* Must be adherent to daily PRO assessments including at least 8 of 14 symptom assessments in the 14 days prior to randomization
* If on background medications for EG/EGE, the medications should be stable at least 4 weeks prior to the run-in period.
* Willing and able to comply with all study procedures and visit schedule including follow-up visits
* Women of childbearing potential must agree to use a highly effective form of birth control (confirmed by the Investigator) from randomization throughout the study duration and within 12 weeks after last dose if IP.

Exclusion criteria:

* Other gastrointestinal disorders such as active Helicobacter pylori infection, history of achalasia, esophageal varices, Crohn's disease, ulcerative colitis, inflammatory bowel disease, or celiac disease.
* Hypereosinophilic syndrome or eosinophilic granulomatosis with polyangiitis.
* Current malignancy, or history of malignancy, except for patients who have had basal cell, localized squamous cell carcinoma of the skin, or in situ carcinoma of the cervix are eligible provided that the patient is in remission and curative therapy was completed at least 12 months prior to the date of informed consent.
* History of anaphylaxis to any biologic therapy or vaccine.
* Current active liver disease.
* Helminth parasitic infection diagnosed within 24 weeks prior to the date informed that has not been treated with or has failed to respond to standard of care therapy.
* Known immunodeficiency disorder including testing positive for HIV.
* Concomitant use of immunosuppressive medication.
* Receipt of live attenuated vaccines 30 days prior to date of informed consent or assent.
* Receipt of inactive vaccines within 7 days of informed consent or assent.
* Initiation or change of a food-elimination diet regimen or re-introduction of a previously eliminated food group from 6 weeks prior to start of the run-in period and unable or unwilling to remain on a stable diet until the completion of Part A and C.
* Currently pregnant or breast-feeding.

Ages: 12 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2024-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc E. Rothenberg, MD, PhD, Principal Investigator — Cincinnati Children's Hospital Medical Center 3333 Burnet Ave, Cincinnati Ohio 45229, United States
Locations (19):
- United States (6):
  - Research Site, Chicago, Illinois
  - Research Site, Boston, Massachusetts
  - Research Site, Rochester, Minnesota
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Salt Lake City, Utah
- Research Site, São Paulo, Brazil
- Italy (3):
  - Research Site, Milan
  - Research Site, Padua
  - Research Site, Pisa
- Japan (4):
  - Research Site, Bunkyō City
  - Research Site, Maebashi
  - Research Site, Ogaki-shi
  - Research Site, Shinjuku-ku
- Research Site, Amsterdam, Netherlands
- Research Site, Staszów, Poland
- Research Site, Seville, Spain
- Research Site, Kyiv, Ukraine
- Research Site, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymised individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de- identified individual patient-level data in an approved sponsor tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: 909_HUDSON_Poster_non-US.pdf — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3258C00001&attachmentIdentifier=04cf3d75-047c-4d62-bcdb-c5fe56049f0a&fileName=909_HUDSON_Poster_non-US.pdf&versionIdentifier=
- See also: 909_HUDSON_Poster_US-enUS.pdf — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3258C00001&attachmentIdentifier=1cb3d679-cf8b-4fd8-9ffa-03db35818d6f&fileName=909_HUDSON_Poster_US-enUS.pdf&versionIdentifier=
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3258C00001&attachmentIdentifier=bc718d03-0e06-45ba-b465-809e811c81a1&fileName=d3258c00001-study-synopsis-ed-1_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 34 participants were screened. Of those, 12 participants were randomised to either the treatment (6 participants) or placebo (participants) arms of the double-blinded treatment period.
Pre-assignment Details: All participants complete a 4-week to 8-week run-in period during which inclusion/exclusion criteria was assessed.
Groups:
- Benralizumab: Patients received benralizumab 30mg every 4 weeks for the 24 weeks treatment period
- Placebo: Patients received matching Placebo every 4 weeks for the 24 weeks treatment period
Period: Double Blind Period
Arm/Group | Benralizumab | Placebo
Started | 6 | 6
Completed | 6 | 3
Not Completed | 0 | 3
Period: Open Label Extension
Arm/Group | Benralizumab | Placebo
Started (All patients (treatment group and placebo group) received benralizumab 30mg every 4 weeks in the open label extension period.) | 6 | 3
Completed | 5 | 2
Not Completed | 1 | 1
Not completed — Subjects who discontinued treatment with study drug in OLE but completed study follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Benralizumab | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 1 | 5 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With a Histologic Response at Week 24
Description: the proportion of patients achieving a histological response at Week 24, is defined as below:
  * 6 eosinophils/hpf in the stomach for the patients with only gastric disease at baseline.
  * 6 eosinophils/hpf in the stomach and ≤15 eosinophils/hpf in the duodenum for the patients with gastric + duodenal disease at baseline.
  * 15 eosinophils/hpf in the duodenum for the patients with only duodenal disease at baseline.
Time Frame: at week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 6 | 6
Participants | 5 | 0

2. Primary Outcome: Change From Baseline in SAGED Score at Week 24
Description: The Symptom Assessment for Gastrointestinal Eosinophilic Diseases (SAGED) instrument was developed to measure gastrointestinal symptoms in participants diagnosed with EG/EGE. It is a daily diary completed by participants each evening from screening until week 76 to record symptoms during the past 24 hours. Severity for each concept is assessed using an 11-point numerical rating scale (0 = 'none' and 10 = 'worst imaginable'). The total SAGED score (range 0-50) is calculated as a 14-day mean of the sum of individual severity items of abdominal pain, nausea, bloating, early satiety and loss of appetite daily. Higher scores indicate greater symptom severity. Three additional items are collected that aren't part of the total SAGED score and are considered separately: severity of vomiting, severity of diarrhoea and frequency of vomiting. Change in SAGED score at week 24 is the week 24 score (study days 155 to 168) minus the baseline score (study days -14 to -1).
Time Frame: at week 24
Measure: Mean (Standard Error); unit: score
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 5 | 3
score | -9.59 (7.26) | -13.69 (4.37)

ADVERSE EVENTS:
Time Frame: AEs in the on-study period are defined as those with onset between day of first dose of study treatment and the day of the scheduled follow-up visit, inclusive, approximately up to Week 88.
Description: Benralizumab = All patients who received benralizumab 30mg every 4 weeks in the double-blind period.
  Placebo= All patients received matching Placebo every 4 weeks in the double-blind period.
  Open Label Benralizumab= All patients received benralizumab 30mg every 4 weeks during the open-label extension period.
Groups:
- Open Label Benralizumab: Patients received benralizumab 30mg every 4 weeks during the open-label extension period.
Arm/Group | Benralizumab | Placebo | Open Label Benralizumab
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/9
Other Adverse Events (participants affected / at risk) | 6/6 | 3/6 | 6/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benralizumab (N=6) | Placebo (N=6) | Open Label Benralizumab (N=9)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Genitourinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sialoadenitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Eating disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Menstrual discomfort (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Myopic chorioretinal degeneration (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to early termination of study limited numbers of patients was randomized and thus data not analysed on group level.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/09/NCT05251909/Prot_008.pdf
  • Statistical Analysis Plan (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/09/NCT05251909/SAP_009.pdf